CLINICAL TRIAL: NCT04704089
Title: Colorimetric Comparison of Email Defects Using Spectrophotometric and Computer Techniques and Biological, Structural and Physico-chemical Analyses of Teeth or Pathological Enamel
Brief Title: Colorimetric, Ultra-structural and Elemental Comparison of Dental Enamel Defects
Acronym: COLOEMAIL
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190001
Record Dates: First submitted 2020-12-18; First posted 2021-01-11 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Amelogenesis Imperfecta; Dental Fluoroses; Hypomineralization Molar Incisor
Keywords: Colorimetry (MeSH); Amelogenesis Imperfecta (MeSH); Dental Fluorosis (MeSH); Molar-incisor-Hypomineralization (MeSH); Developmental Enamel Defects (MeSH); Shade selection; Dental color matching; Diagnosis (MeSH)
MeSH Terms: conditions — Amelogenesis Imperfecta; Fluorosis, Dental; Molar Hypomineralization; Developmental Defects of Enamel; Disease | interventions — Biological Products; Microscopy, Electron

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- spectrophotometer, and numerical values of tooth color in the populations studied: at the first visit Shooting with Spectrophotometer and at the second visit for all patients except control population: Tooth extraction or restorative treatment Collection of teeth or enamel debris for analysis
  Interventions: Other: spectrophotometer; Other: Biological (protein analysis by western blot or mass spectrometry of matrix proteins), structural (electron microscopy) and physico-chemical analyses

INTERVENTIONS:
Other: spectrophotometer — * Calibration of the spectrophotometer (calibration of white and green color on the provided support),
  * Placing the patient or witness in the chair,
  * Placement of intraoral retractors,
  * Photographs of the dental arch in occlusion as well as slightly open mouth to visualize the mandibular incisors,
  * If MIH is suspected, occlusal images of the occlusal surfaces of the first molars will be taken with the help of a dental mirror,
  * Shooting with the spectrophotometer centered on each of the teeth of interest in the anterior sector with verification of the good quality of the shot according to the axis (validated in green on the camera),
  * Backup of images with coded identification number
Other: Biological (protein analysis by western blot or mass spectrometry of matrix proteins), structural (electron microscopy) and physico-chemical analyses — * Chemical analysis of enamel mineral.
  * Techniques of spectrometry and spectroscopy (Raman and FTIR)
  * Atomic Probe Tomography and Protein Mass Spectrometry (ICP-MS).

SUMMARY:
The study focuses on the analysis of enamel defects grouping together hypomineralization and hypoplasia. It focuses on 3 very characteristic enamel pathologies that are most often encountered in dental consultations: Molar Incisor Hypomineralization (MIH), dental fluorosis (FD) and amelogenesis imperfecta (AI). The research focuses on the use of a spectrophotometer for measuring tooth colors: the Zfx SpectroShade® (MHT) and its software as a means of early diagnosis of pre-eruptive enamel abnormalities. The main objective of the study is to analyze the color parameters of teeth affected with one of the 3 enamel abnormalities for use of the spectrophotometer as a non-invasive diagnostic tool for enamel defects.

The secondary objective is focused on the biological, structural and physicochemical characterizations of these different enamel pathologies from extracted teeth or enamel biopsies that must be ground to achieve a restoration.

DETAILED DESCRIPTION:
Methodology:

V1 inclusion visit (D1):

The subjects will be screened during a consultation carried out as part of the treatment in the participating dentistry departments. The inclusion and non-inclusion criteria for participants will be verified and the study will be offered to eligible patients and controls. The research briefing note will be given and the non-objection of the participants (adults and representative (s) of parental authority) will be collected. The investigator will then take the photographs and spectrophotometer shots (at least 2 teeth per participant).

V2 follow-up visit (within 2 months of the inclusion visit (D2 to M2)):

The patients will be reviewed in consultation as part of the treatment for selective grinding for dental restoration or extraction (if the tooth (s) is (are) no longer storable). The teeth or pathological enamel samples will be recovered and centralized at the Laboratory of Oral Molecular Physiopathology.

Biological, structural and physico-chemical analyzes will be carried out from these samples.

In order to ensure follow-up of participants, the principal investigator of each center will maintain a correspondence table including the participant's identity and his research identification number. He will also keep a register of oppositions up to date.

The subject's opposition or participation will be notified in his medical file. A copy of the briefing notes and non-objection forms signed by the dentist will be kept on site with the research documents. Minors who become adults during their participation will benefit from appropriate information and their non-objection will be collected.

Primary endpoint Analysis, using the spectrophotometer, of the numerical values of the color of the teeth in each of the populations studied (Hereditary amelogenesis imperfecta (AIH), dental fluorosis (FD), Hypomineralization Incisors and Molar (MIH) and control).

For each pathology, the values of these parameters will be compared. Secondary endpoints

* Intra-pathology classification according to the severity of each pathology.
* Characterization and biological, structural and physicochemical analysis of these different pathologies from extracted teeth or enamel biopsy to be ground to achieve a restoration.

Sample analysis The teeth samples will be stored at room temperature in the Oral Molecular Physiopathology laboratory in the Research Center.

During the research, biological, structural and physicochemical analyzes will be carried out at the laboratory or in another laboratory in France or abroad. A contract will be established upstream of these analyzes with the partner laboratory.

At the end of the research, samples not destroyed by destructive analysis techniques will be embedded in the resin and stored for 10 years before being destroyed. These samples can be used for additional analyzes (biological, structural and physico-chemical) according to the request of the references for the publication process.

ELIGIBILITY:
For patients :

Inclusion Criteria :

1. Age between 8 and 55 years old
2. Carrier of one of the following 3 quantitative pre-eruptive enamel anomalies : AIH, dental fluorosis or MIH
3. Information and collection of the non-opposition of the adult patient or of the representative(s) of parental authority present for the minors.

Criteria for non-inclusion :

1. Pregnant or breastfeeding woman
2. Under guardianship or curators
3. Opposition of the minor patient
4. Presenting pre-eruptive anomalies only on the molars (the spectrophotometer can only take pictures of the anterior dental sector (incisors and canines)).
5. Other types of hypomineralization (post-eruptive, of traumatic or infectious origin, idiopathic).
6. Having undergone radiotherapy or chemotherapy inducing dental and periodontal damage.
7. Having systemic abnormalities (unbalanced diseases), haemochromatosis, porphyria
8. Under medication likely to disturb the coloring of the teeth

For witnesses :

Inclusion Criteria :

1. Age between 8 and 55 years old
2. Information and collection of the non-opposition of the adult witness or of the representative(s) of parental authority present for the minors.
3. Free of any anomaly of tooth structure, exogenous dyschromia and carious lesions.

Criteria for non-inclusion :

1. Pregnant or breastfeeding woman
2. Under guardianship or curators
3. Opposition of the minor witness
4. Carrier of a quantitative pre-eruptive enamel anomaly
5. Polycarpus (preventing the diagnosis of amyl hypomineralization)

Ages: 8 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Major or minor patients with Hereditary Imperfect Amelogenesis Imperfecta (HIA), Dental Fluorosis (DF), Incisor and Molar Hypomineralization (MIH) or Control
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2026-04-18 (Estimated)

PRIMARY OUTCOMES:
analyze the color parameters of teeth presenting one of the 3 enamel anomalies in order to use the spectrophotometer as a non-invasive diagnostic tool for enamel dyschromia. | at the first visit = inclusion visit

SECONDARY OUTCOMES:
Biological characterization of the proteins of the dental enamel matrix by Western Blot and/or mass spectrometry from samples (extracted teeth or enamel biopsies to be ground during the treatment). | at the second visit, 2 months after inclusion visit and after tooth extraction
Ultra-structural characterization under electron microscope and biomechanics by nanoindentation of enamel pathologies from extracted teeth or enamel biopsies to be ground during the treatment. | at the second visit, 2 months after inclusion visit and after tooth extraction
Physico-chemical characterization by different spectroscopic techniques of enamel pathologies from extracted teeth or enamel biopsies to be ground during the treatment. | at the second visit, 2 months after inclusion visit and after tooth extraction
Physico-chemical characterization by atomic probe tomography of enamel pathologies from extracted teeth or enamel biopsies to be ground during the treatment. | at the second visit, 2 months after inclusion visit and after tooth extraction

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'odontologie, Hôpital Pitié-Salpêtrière, Paris, France